CLINICAL TRIAL: NCT02703818
Title: Multi-Center, Prospective, Clinical Trial of the Senza™ Spinal Cord Stimulation (SCS) System in the Treatment Of Chronic Pain of the Upper Extremities
Brief Title: SCS for the Treatment Of Chronic Pain of the Upper Extremities
Acronym: UEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nevro Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA2015-4 US
Record Dates: First submitted 2016-03-02; First posted 2016-03-09 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Upper Extremity Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Senza (Experimental): Spinal Cord Stimulation for UEP
  Interventions: Device: Senza

INTERVENTIONS:
Device: Senza — Spinal Cord Stimulation

SUMMARY:
This is a prospective, multi-center post-market study of the Senza System in subjects with chronic, intractable pain of the upper extremities. Data at follow-up visits will be compared to Baseline data collected at the beginning of the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Have been diagnosed with chronic, intractable pain of an upper extremity of neuropathic origin, which has been refractory to conservative therapy for a minimum of 3 months.
2. Have an average pain intensity (over a period of 7 days) of an upper extremity of ≥ 5 out of 10 cm on the Visual Analog Scale (VAS) at enrollment.
3. Be on stable pain medications for at least 28 days and be willing to stay on those medications with no dose adjustments until activation of the permanently implanted SCS device.
4. Be 18 years of age or older at the time of enrollment.
5. Be an appropriate candidate for the surgical procedures required in this study.
6. Be capable of subjective evaluation, able to read and understand English-written questionnaires, and are able to read, understand and sign the written inform consent in English.
7. Have stable neurological status measured by motor, sensory and reflex function.

Key Exclusion Criteria:

1. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures.
2. Have a current diagnosis of a progressive neurological disease.
3. Have a current diagnosis or condition such as a coagulation disorder, bleeding diathesis, platelet dysfunction, progressive peripheral vascular disease or uncontrolled diabetes mellitus that presents excess risk for performing the procedure.
4. Have mechanical spine instability as determined.
5. Have significant stenosis, based on MRI.
6. Have an existing drug pump and/or another active implantable device (switched on or off) such as a pacemaker or other SCS devices.
7. Have a condition currently requiring or likely to require the use of whole body MRI or diathermy.
8. Be pregnant (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile or be at least 2 years post-menopausal).
9. Have within 6 months of enrollment a significant untreated addiction to dependency producing medications, alcohol or illicit drugs.
10. Be involved in an injury claim under current litigation.
11. Have a pending or approved worker's compensation claim.
12. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention and/or ability to evaluate treatment outcome, as determined by a psychologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Responder Rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: David Caraway, MD, Study Director — Nevro Corp
Locations (1):
- NEVRO Corp, Redwood City, California, United States

REFERENCES:
- [Derived] Burgher A, Kosek P, Surrett S, Rosen SM, Bromberg T, Gulve A, Kansal A, Wu P, McRoberts WP, Udeshi A, Esposito M, Gliner BE, Maneshi M, Rotte A, Subbaroyan J. Ten kilohertz SCS for Treatment of Chronic Upper Extremity Pain (UEP): Results from Prospective Observational Study. J Pain Res. 2020 Nov 10;13:2837-2851. doi: 10.2147/JPR.S278661. eCollection 2020. PMID 33204145